CLINICAL TRIAL: NCT03861624
Title: Intramedullary Nailing Versus External Fixation in the Treatment of Open Tibia Fractures in Tanzania - Results of a Randomized Controlled Trial
Brief Title: Intramedullary Nailing Versus External Fixation in Open Tibia Fractures in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Wyss Foundation, Inc (Unknown); Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-14792
Record Dates: First submitted 2019-02-25; First posted 2019-03-04 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Tibial Fractures; Open Fracture of Tibia; Trauma
Keywords: Tibia; Intramedullary nailing; External fixation; Trauma
MeSH Terms: conditions — Tibial Fractures; Wounds and Injuries | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intramedullary nailing (Experimental): Patients receive definitive fixation of AO/OTA-42 open tibia diaphyseal fractures via Intramedullary nailing with standard SIGN nail.
  Interventions: Procedure: Intramedullary nailing with standard SIGN nail
- External Fixation (Active Comparator): Patients receive definitive fixation of AO/OTA-42 open tibia diaphyseal fractures External Fixation with uniplanar Dispofix external fixator.
  Interventions: Procedure: External Fixation with uniplanar Dispofix external fixator

INTERVENTIONS:
Procedure: Intramedullary nailing with standard SIGN nail — Patients meeting eligibility requirements are randomized to either study arm. Patients receive definitive fixation of AO/OTA-42 open tibia diaphyseal fractures using the standard SIGN nail (SIGN Fracture Care International, Richland, WA). The number of interlocking screws is at the discretion of the treating surgeon, who also has the option to use an external fixator for damage control, and later conversion to IMN when clinically appropriate. The experimental group procedure is less common in the study setting, and thus, viewed as the experimental group.
  Arms: Intramedullary nailing
Procedure: External Fixation with uniplanar Dispofix external fixator — Patients meeting eligibility requirements are randomized to either study arm. Patients receive definitive fixation of AO/OTA-42 open tibia diaphyseal fractures using the uniplanar Dispofix external fixator with two Shanz screws placed proximally and two Schanz screws placed distally to fracture site with a single stainless steel bar.The active comparator group procedure is more common in the study setting, and thus, viewed as the comparator group.
  Arms: External Fixation

SUMMARY:
The investigators propose to undertake a randomized, controlled trial which will generate Level 1 evidence concerning optimal fixation methods for the treatment of severe open tibia fractures in Dar es Salaam, Tanzania. The investigators hope to determine the optimal management of severe open tibial fractures in Sub-Saharan Africa in order to reduce long-term disability, limit the economic impact of injury, and avoid resource costs of reoperation. The investigators plan to compare the all-cause reoperation rate for AO/Orthopaedic Trauma Association (OTA) Type 42 open tibial shaft fractures treated with initial intramedullary nailing versus external fixation at Muhimbili Orthopaedic Institute in Dar es Salaam, Tanzania, to compare rates of secondary clinical endpoints including postoperative superficial and deep infection, clinical union, radiographic union, malunion, and health-related quality of life with minimum one year follow-up, and identify prognostic factors related to the patient, injury, or management protocol that impact the reoperation rate, return to work, and health-related quality of life.

DETAILED DESCRIPTION:
The investigators conducted a prospective randomised controlled trial at a tertiary referral hospital in Dar es Salaam, Tanzania from December 17th, 2015 to March 25th, 2017. All open tibia fractures arriving at the hospital emergency room during the enrollment period were screened for inclusion in the study. Inclusion and exclusion criteria are noted later in this submission.All patients who were eligible after clinical screening were offered enrollment in the study and subsequently completed written informed consent in either English or Swahili depending on the patient's preference. The investigation was approved by ethical review boards at the University of California San Francisco (UCSF) and the Tanzanian National Institute for Medical Research (NIMR).

All enrolled participants were taken to the operating room for initial irrigation and debridement using a standardized protocol aiming for debridement within 24 hours of hospital admission. Preoperative ceftriaxone was given as soon as possible after presentation to the emergency department. Following debridement, the primary surgeon determined if the wound was amenable to immediate or delayed primary closure. If amenable to primary closure, the patient was randomized by a site research coordinator to one of two treatments (Intramedullary nailing (IMN) or external fixation (EF))using a centralized web-based electronic randomization tool, Research Electronic Data Capture (REDCap). The study computer analyst developed the REDCap randomization module with input from senior authors. The REDCap randomization module incorporated block randomization to maintain equal patient distribution between each treatment group and to ensure allocation concealment.

Data from a pilot study at the site of our investigation informed sample size calculations, which showed reoperation rates of external fixation and intramedullary nailing of 38% versus 3.8%. However, with longer follow-up and more stringent criteria for a primary event, The investigators used a more conservative effect size of 20% compared to 5%. Using a power of 80% and alpha of 0.05, The investigators calculated the study would require 88 patients in each treatment group (176 total). Accounting for 20% loss to follow up, The investigators estimated a total sample size requirement of 240 patients (120 per group).

Data monitoring was completed by the adjudication committee at 6 month intervals throughout the study duration and prior to final analysis in December, 2018.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletal maturity
2. AO/OTA 42 open tibia fractures
3. Wound primarily closeable (no flap or delay in closure due to contamination needed)
4. Palpable pedal pulses (no vascular injury sustained)
5. Presentation within 24 hours from injury

Exclusion Criteria:

1. Current injury is a pathologic fracture
2. Sustained bilateral tibia fracture
3. Sustained comminuted femur fracture
4. Sustained severe Traumatic Brain Injury (GCS<12) ***
5. Sustained severe spinal cord injury (lower extremity paresis/paralysis)
6. Sustained severe burns (>10% total body surface area (TBSA) or >5% TBSA with full thickness or circumferential injury)
7. Prior ipsilateral leg injury requiring surgery
8. Prior or current lower limb deformity or abnormality
9. Unable to complete follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2017-03-25 (Actual); Study Completion 2017-03-25 (Actual)

PRIMARY OUTCOMES:
Rate of composite, all-cause reoperation | One year of definitive skeletal stabilization
  The use of composite outcomes has been validated in a wide range of clinical trials. Primary events included in the composite outcome include: infection or hematoma, bone grafting, implant conversion or exchange >6 weeks after index procedure, implant removal, dynamization of intramedullary nail, osteotomy, amputation.

SECONDARY OUTCOMES:
Rate of superficial infection | Assessed at clinical follow-up appointments at 2, 6, 12, 26, and 52 weeks
  As defined by center for disease control (CDC) surveillance definitions, to include pin tract infections and cellulitis which resolves with use of antibiotics and local wound care.
Rate of deep infection | Assessed at clinical follow-up appointments at 2, 6, 12, 26, and 52 weeks
  As defined by CDC surveillance definitions, to include deep abscess or osteomyelitis.
Number of participants with clinical nonunion | Assessed at clinical follow-up appointments at 6, 12, 26, and 52 weeks
  Union of fracture healing will be assessed by absence of movement at fracture site and time to painless weight bearing. Non-union will be defined as fracture failure to heal beyond six months from date of injury.
Number of participants with radiographic nonunion | Assessed at clinical follow-up appointments at 6, 12, 26, and 52 weeks
  Radiographic union will be assessed using rate of callous formation and visibility of fracture line as measured by the Radiographic union score for tibia (RUST) score
Number of participants with malunion | Assessed at clinical follow-up appointments at 6, 12, 26, and 52 weeks
  Post-operative malalignment will be defined as leg length discrepancy (>1 cm shortening), angular malalignment (> 5 degrees sagittal or coronal angulation referenced contralateral leg radiographs, if non-injured), or malrotation (>10 degrees, determined by Foot-Thigh Angle).
Number of participants with implant failure | Assessed at clinical follow-up appointments at 2, 6, 12, 26, and 52 weeks
  Implant failure will be defined as breakage or loosening of any implant component at bone-implant interface which necessitates re-operation.
Health-related quality of life | Assessed at 2, 6, 12, 26, and 52 week time point.
  Health related quality of life measured by Euro Quality of Life-5 Dimension (EuroQoL-5D, EQ5D) Index.
  Contains 5 domains: Mobility, Self-Care, Usual activities, Pain/discomfort, Anxiety/depression Each domain contains 3 levels of health state pertaining to that level. Index score is calculated via weighted scores across each domain. Measured from 0 to 1 where 0 is equivalent to death and 1 is equivalent to perfect state of health.
Visual analogue pain score | Assessed at 2, 6, 12, 26, and 52 week time point.
  Visual analogue pain score represents a patient's current level of pain scored from 1-10 where 1 = no/minimal pain to 10 = worst possible pain.
Participant knee range of motion | Assessed at 6, 12, 26, and 52 week time point.
  Includes:
  * Maximum knee extension/flexion as measured with a goniometer
  * Values are recorded in degrees from neutral/hyperextension to ≥ 30 by intervals of 5 degrees for maximum knee extension
  * Values are recorded in degrees from ≤30 degrees to ≥140 degrees by intervals of 10 degrees for maximum knee flexion
Participant ankle range of motion | Assessed at 6, 12, 26, and 52 week time point.
  Includes:
  * Maximum ankle dorsiflexion/plantarflexion as measured with a goniometer
  * Values are recorded in degrees from -15 degrees to >25 degrees by intervals of 5 degrees for maximum ankle dorsiflexion
  * Values are recorded in degrees from <10 degrees to >50 degrees by intervals of 10 degrees for maximum ankle plantarflexion
Participant ability to perform Squat and Smile test | Assessed at 6, 12, 26, and 52 week time point.
  The Squat and Smile test (S&S) is a functional assessment of squatting ability used by SIGN Fracture Care International to quickly assess fracture healing.
  Squat depth is categorized by squat level: unable (1), above knee level (2), at knee level (3) or below knee level (4)
  -Values are scored from 1 to 4 where 1 is worst and 4 is best.
  Support component is categorized by: requiring both hands for support with squatting (1), one hand for support with squatting (2), or no hands for support with squatting (3) -Values are scored from 1 to 3 where 1 is worst and 3 is best
  Smile component is categorized into painful grimace (1), neutral expression (2), and smile (3) where painful grimace is worst and smile is best.
  -Values are scored from 1 to 3 where 1 is worst and 3 is best
  Each component is scored and evaluated individually as separate domains. There is no pooling of scores.
Patient speed in completing walking speed test according to NIH 4 meter walking test | Assessed at 6, 12, 26, and 52 week time point.
  Measures locomotion
  Participants walk 4 meters at their usual pace and complete one practice and two timed trials. Raw scores are recorded at the time in seconds required to walk four meters on each of the two trials with the better trial used as the final score.

CONTACTS AND LOCATIONS:
Overall Officials: Saam Morshed, MD, MPH, Study Chair — University of California, San Francisco; David Shearer, MD, MPH, Principal Investigator — University of California, San Francisco; Billy Haonga, MD, Principal Investigator — Muhimbili Orthopaedic Institute; Edmund Eliezer, MD, Principal Investigator — Muhimbili Orthopaedic Institute

IPD SHARING:
Plan to Share IPD: Yes
The data for this study including deidentified participant data and a data dictionary will be made available upon request. The study protocol, statistical analysis plan, and informed consent forms will also be made available upon request. These data and documents will be available with publication. Data and document access can be granted through email correspondence with the corresponding author and will require a signed data access agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available upon publication. There is no expiration period for data availability.
Access Criteria: Investigators requesting data access will be required to submit a cover letter and email to the primary study contact outlining their reasons for requesting data access and their plan for use of study data. All decisions to allow access will be determined by study principal investigators.

REFERENCES:
- [Background] Chandran A, Hyder AA, Peek-Asa C. The global burden of unintentional injuries and an agenda for progress. Epidemiol Rev. 2010;32(1):110-20. doi: 10.1093/epirev/mxq009. Epub 2010 Jun 22. PMID 20570956
- [Background] Patton GC, Coffey C, Sawyer SM, Viner RM, Haller DM, Bose K, Vos T, Ferguson J, Mathers CD. Global patterns of mortality in young people: a systematic analysis of population health data. Lancet. 2009 Sep 12;374(9693):881-92. doi: 10.1016/S0140-6736(09)60741-8. PMID 19748397
- [Background] Mock C, Cherian MN. The global burden of musculoskeletal injuries: challenges and solutions. Clin Orthop Relat Res. 2008 Oct;466(10):2306-16. doi: 10.1007/s11999-008-0416-z. Epub 2008 Aug 5. PMID 18679760
- [Background] Beveridge M, Howard A. The burden of orthopaedic disease in developing countries. J Bone Joint Surg Am. 2004 Aug;86(8):1819-22. doi: 10.2106/00004623-200408000-00029. PMID 15292432
- [Background] WHO Scientific Group on the Burden of Musculoskeletal Conditions at the Start of the New Millennium. The burden of musculoskeletal conditions at the start of the new millennium. World Health Organ Tech Rep Ser. 2003;919:i-x, 1-218, back cover. PMID 14679827
- [Background] Dormans JP, Fisher RC, Pill SG. Orthopaedics in the developing world: present and future concerns. J Am Acad Orthop Surg. 2001 Sep-Oct;9(5):289-96. doi: 10.5435/00124635-200109000-00002. PMID 11575908
- [Background] Museru LM, Mcharo CN. The dilemma of fracture treatment in developing countries. Int Orthop. 2002;26(6):324-7. doi: 10.1007/s00264-002-0408-7. Epub 2002 Oct 17. No abstract available. PMID 12466862
- [Background] Zirkle LG Jr. Injuries in developing countries--how can we help? The role of orthopaedic surgeons. Clin Orthop Relat Res. 2008 Oct;466(10):2443-50. doi: 10.1007/s11999-008-0387-0. Epub 2008 Aug 7. PMID 18685912
- [Background] Shah RK, Moehring HD, Singh RP, Dhakal A. Surgical Implant Generation Network (SIGN) intramedullary nailing of open fractures of the tibia. Int Orthop. 2004 Jun;28(3):163-6. doi: 10.1007/s00264-003-0535-9. Epub 2004 Jan 9. PMID 14714143
- [Background] Shearer D, Cunningham, B., Zirkle, L. Population Characteristics and Clinical Outcomes from the SIGN Online Surgical Database. Techniques in Orthopaedics. 2009;24(4):273-276.
- [Background] Ikpeme I, Ngim N, Udosen A, Onuba O, Enembe O, Bello S. External jig-aided intramedullary interlocking nailing of diaphyseal fractures: experience from a tropical developing centre. Int Orthop. 2011 Jan;35(1):107-11. doi: 10.1007/s00264-009-0949-0. Epub 2010 Feb 11. PMID 20148329
- [Background] Ogunlusi JD, St Rose RS, Davids T. Interlocking nailing without imaging: the challenges of locating distal slots and how to overcome them in SIGN intramedullary nailing. Int Orthop. 2010 Aug;34(6):891-5. doi: 10.1007/s00264-009-0882-2. Epub 2009 Oct 8. PMID 19813011
- [Background] Naeem-Ur-Razaq M, Qasim M, Khan MA, Sahibzada AS, Sultan S. Management outcome of closed femoral shaft fractures by open Surgical Implant Generation Network (SIGN) interlocking nails. J Ayub Med Coll Abbottabad. 2009 Jan-Mar;21(1):21-4. PMID 20364733
- [Background] Ikem IC, Ogunlusi JD, Ine HR. Achieving interlocking nails without using an image intensifier. Int Orthop. 2007 Aug;31(4):487-90. doi: 10.1007/s00264-006-0219-3. Epub 2006 Oct 13. PMID 17039384
- [Background] Sekimpi P, Okike K, Zirkle L, Jawa A. Femoral fracture fixation in developing countries: an evaluation of the Surgical Implant Generation Network (SIGN) intramedullary nail. J Bone Joint Surg Am. 2011 Oct 5;93(19):1811-8. doi: 10.2106/JBJS.J.01322. PMID 22005867
- [Background] Kooistra BW, Dijkman BG, Busse JW, Sprague S, Schemitsch EH, Bhandari M. The radiographic union scale in tibial fractures: reliability and validity. J Orthop Trauma. 2010 Mar;24 Suppl 1:S81-6. doi: 10.1097/BOT.0b013e3181ca3fd1. PMID 20182243

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT03861624/Prot_ICF_000.pdf